CLINICAL TRIAL: NCT05013320
Title: Combined Dexmedetomidine and Glycopyrrolate Therapy for Prevention of Catheter Related Bladder Discomfort After Transurethral Bladder Surgery
Brief Title: Combined Dexmedetomidine and Glycopyrrolate Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not get the IRB approval
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEXLYCO
Record Dates: First submitted 2021-05-13; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Bladder Irritable
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Glycopyrrolate; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine only (Active Comparator): dexmedetomidine is administered during the surgery
  Interventions: Drug: Dexmedetomidine
- Combined dexmedetomidine and glycopyrrolate (Experimental): glycopyrrolate and dexmedetomidine are administered during the surgery
  Interventions: Drug: Glycopyrrolate + dexmedetomidine

INTERVENTIONS:
Drug: Glycopyrrolate + dexmedetomidine — Intravenous glycopyrrolate before anesthetic induction. Dexmedetomidine administration during the surgery.
  Arms: Combined dexmedetomidine and glycopyrrolate
Drug: Dexmedetomidine — Dexmedetomidine administration during the surgery.
  Arms: Dexmedetomidine only

SUMMARY:
Catheter-related bladder discomfort after transurethral resection of bladder tumor is frequent because of indwelling urinary catheter for irrigation. The mechanism of the catheter-related bladder discomfort is similar to that of overactive bladder, in which muscarinic acetylcholine receptors are stimulated. The catheter-related bladder discomfort is a well known predisposing factor for emergence delirium after general anesthesia. In this study, we aimed to compare the incidence of catheter-related bladder discomfort between dexmedetomidine only therapy and combind dexmedetomidine and glycopyrrolate therapy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II
* elective transurethral resection of bladder tumor under general anesthesia

Exclusion Criteria:

* arrhythmia
* bladder outflow obstruction
* overacitve bladder
* end stage renal disease
* neurogenic bladder
* morbid obesity
* psychiatric disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of catheter-related bladder discomfort | 0 minute after entering the post-anesthetic care unit
  No = not complaining of bladder discomfort on asking; Mild = report discomfot only on questioning; Moderate: report without questioning without behavior responses; Severe = report without questioniing accompanied by behavior responses. Mild, Moderate, Severe bladder discomfort is defined to have catheter-related bladder discomfort

SECONDARY OUTCOMES:
Emergence agitation | 0 minute, 30 minute, and 6 hours after entering the post-anesthetic care unit
  (1)calm (2)slightly agitated but consolable (3)moderately agitated and inconsolable (4)severely agitated and highly inconsolable
Delirium | 0 minute, 30 minute, and 6 hours after entering the post-anesthetic care unit
  (1)acute and fluctuating changes in mental status (2)inattention (3)disorganized or incoherent thinking (4)altered level of consciousness. (1),(2) and (3), (1),(2), and (4), or (1)(2)(3)and (4) are defined to have deilrium.
Postoperative pain | 0 minute, 30 minute, and 6 hours after entering the post-anesthetic care unit
  numerical rating scale (0=no pain to 10=worst pain imaginable)
Sedation score | 0 minute, 30 minute, and 6 hours after entering the post-anesthetic care unit
  (1)anxious, agitated or restless (2)cooperative, oriented and trranquil (3)responds to commands, asleep (4)brisk response to light glabellar taps or oud noise (5)sluggish response to light glabellar taps or loud noise (6)noresponse
Dry mouth | 0 minute, 30 minute, and 6 hours after entering the post-anesthetic care unit
  yes or no
postoperative nausea and vomiting | 0 minute, 30 minute, and 6 hours after entering the post-anesthetic care unit
  yes or no